CLINICAL TRIAL: NCT04235283
Title: Comparison of the Radiographic Outcomes and Total Blood Loss Between Pinless Navigation and Conventional Method in Minimally Invasive Total Knee Arthroplasty
Brief Title: Comparison of Pinless Navigation and Conventional Method in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMRPG8J0311
Record Dates: First submitted 2020-01-17; First posted 2020-01-21 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Total knee arthroplasty; pinless; navigation; alignment; minimal invasive
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Enroll 100 patients who plan to undergo unilateral primary MIS-TKA and will be randomly assigned into two groups. The first group (50 patients) will be treated by pinless-navigation (Stryker, OrthoMap Express Knee Navigation) MIS-TKA, and the second group (50 patients) will undergo traditional MIS-TKA.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study proposed 1:1 randomization into pinless navigation and conventional technique. Each patient who enrolled in this study will be given sequence study number, and the chief surgeon will draw lots to decide which group will be assigned in. The patient and the independent reviewer are kept blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group I (Experimental): Primary total knee replacement by pinless navigation and minimally invasive technique
  Interventions: Device: Primary total knee replacement by pinless navigation (Orthomap Express,Stryker, Michigan)
- Group II (Active Comparator): Primary total knee replacement by traditional jig and minimally invasive technique
  Interventions: Procedure: Primary total knee replacement by traditional jig and minimally invasive technique

INTERVENTIONS:
Device: Primary total knee replacement by pinless navigation (Orthomap Express,Stryker, Michigan) — The varus/valgus, extension/flexion, thickness of distal cut of femur was determined and done by pinless navigation system. After cutting, the instant information of resection level can show on the display screen. If the alignment is satisfying, the anterior/posterior femoral cut, chamfer cut and box resection were done by conventional jig
  Arms: Group I
Procedure: Primary total knee replacement by traditional jig and minimally invasive technique — The femoral alignment was determined by intramedullary guide. The femoral alignment jig was set to 5-7 degree valgus dependent on the preoperative radiograph. A bone plug is impacted into the entry hole of femoral medullary canal before prosthesis placement.
  Arms: Group II

SUMMARY:
The purpose of this study is to conduct a prospective randomized clinical trial to compare the accuracy of prosthesis, radiographic alignment, total blood loss, the risk of venous thromboembolism between pinless-navigated total knee arthroplasty (TKA) and traditional TKA.

DETAILED DESCRIPTION:
Minimal invasive surgery total knee arthroplasty (MIS-TKA) is an excellent surgical procedure for patients with end-stage knee diseases and can reduce the postoperative complications compared with traditional TKA procedures.

However, MIS-TKA procedures require a long learning curve to avoid malposition of prosthesis. In previous studies have demonstrated that the position of prosthesis and the postoperative mechanical axis are critical factors of outcome. Malposition of prosthesis and deviation more than 3 degrees of mechanical axis will lead to asymmetrical tibia-femoral tracking between prosthesis with the wear of linear, and increase the incidence of prosthesis loosening.

Computer navigation assisted system has been used in TKA procedures for more than one decade and has been proven to improve the accuracy of prosthesis placement and postoperative mechanical alignment. Moreover, navigated TKA avoids the use of intramedullary guide and preserve the medullary cavity of femur, so the risks of bleeding and venous thromboembolism are reduced. However, traditional navigation system requires additional procedure to set reference arrays with pin fixation of femur and tibia. Pin wound complications including bleeding, infection, and iatrogenic fracture were reported. Moreover, traditional navigation system requires conventional TKA approach in which the wound length of the knee will be as long as 15 to 20 cm. Therefore a combination of new navigation system with a MIS technique to perform TKA procedure is required The new pinless navigated system for TKA procedures has been developed, as the navigation tools were fixed in the surgical field without additional pin wounds. This advantage meets the rationale of MIS-TKA to take care of both minimal invasive procedures and accuracy of prosthesis placement. Therefore, the investigators want to investigate the application of this pinless navigation system in MIS-TKA procedures.

Our purpose is to conduct a prospective randomized clinical trial to compare the accuracy of prosthesis, radiographic alignment, total blood loss, the risk of venous thromboembolism between pinless-navigated MIS-TKA and traditional MIS-TKA.

Material and Methods:

The investigators plan to enroll 100 patients who plan to undergo unilateral primary MIS-TKA and will be randomly assigned into two groups. The first group (50 patients) will be treated by pinless-navigation (Stryker, OrthoMap Express Knee Navigation) MIS-TKA, and the second group (50 patients) will undergo traditional MIS-TKA.

The investigators will record the surgical wound length, surgical time cost and calculate daily hemoglobin drainage and total blood loss after TKA procedures for all patients. At 3 months after operation, the whole leg scanography, AP and lat view of knee radiography will be take and the mechanical alignment (MA), anatomic alignment (AA), femoral bowing angle (FBA), and coronal femoral-component angle (CFA), coronal tibia-component angle (CTA) in coronary view and sagittal femoral component angle (SFA), sagittal tibial component angle (STA) in lateral view will be measured. The operating time and surgical wound length in knee full extension will be recorded. All complications including bleedings, wound complications, venous thromboembolism will be recorded.

Study year: one year Expecting Result The investigators anticipate that the position of prosthesis in pinless-navigated MIS-TKA is more accurate or equal to traditional MIS-TKA group. And the total blood loss in pinless-navigated MIS-TKA is less than traditional MIS-TKA group. The complication rate is similar between the two groups

ELIGIBILITY:
Inclusion Criteria:

1. Patients with osteoarthritis of the knee secondary to degeneration, inflammatory arthritis, gouty arthritis, posttraumatic arthritis, and undergoing primary unilateral minimally invasive TKA
2. Age > 50 years and < 90 years
3. Failure of medical treatment or rehabilitation.
4. Hemoglobin > 11g/dl,
5. No use of non-steroid anti-inflammatory agent one week before operation

Exclusion Criteria:

1. Preoperative Hemoglobin <11 g/dl
2. History of infection or intraarticular fracture of the affective knee
3. Renal function deficiency (GFR <30 ml/min/1.73m2)
4. Elevated liver enzyme (AST/ALT level are more than twice normal range) , history of liver cirrhosis, impaired liver function(elevated total bilirubin level) and coagulopathy (including long-term use anticoagulant)
5. History of deep vein thrombosis, ischemic heart disease, cardiac arrythmia requiring life-long anti-coagulants, or stroke
6. Contraindications of tranexamic acid, rivaroxaban, or the excipients
7. Allergy to tranexamic acid, rivaroxaban, or the excipients
8. Coagulopathy or bleeding tendency caused by organ dysfunction, such as cirrhosis, bone marrow suppression etc.
9. Patient who have active bleeding disorder, such as intracranial hemorrhage, upper GI bleeding, hematuria

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic outcome: the mechanical alignment (MA) | Three months after operation
  The mechanical alignment (MA): an angle between the mechanical axis of the femur and the tibial shaft axis
Radiographic outcome: anatomic alignment (AA) | Three months after operation
  The anatomic alignment (AA): an angle between the axis of the femoral shaft and the tibial shaft axis
Radiographic outcome: femoral bowing angle (FBA) | Three months after operation
  The femoral bowing angle (FBA): the angle between the distal and proximal femoral anatomical axes
Radiographic outcome: coronal femoral-component angle (CFA) | Three months after operation
  Tthe angle between the femoral mechanical axis and the femoral component
Radiographic outcome: coronal tibia-component angle (CTA) | Three months after operation
  The angle between the tibial shaft axis and the tibial component

SECONDARY OUTCOMES:
Total Blood Loss | Postoperative Day 3
  The total blood loss was calculated according to Nadler et al., which uses maximum postoperative decrease of the Hb level adjusted for weight and height of the patient. Total blood loss consists of amount of blood loss calculated from the maximum Hb loss and amount of blood transfused
Blood transfusion rate | Three months after operation
  Record the event of blood transfusion, and calculate the incidence of transfusion
Operating Time | After the procedure is done
  Time needed for the surgical procedure (skin to skin) is recorded
Surgical wound length | After the procedure is done
  The surgical wound length at full extension of knee is also recorded
Wound complications | Three months after operation
  Any wound complications including superficial infection, wound dehiscence, poor healing, etc. are all recorded
Venous thromboembolism | Postoperative Day 4
  perform duplex ultrasound study of both lower limbs in all patients on postoperative day 4

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Wen Wang, MD, Study Director — Department of Orthopaedic Surgery, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang Z, Zhu W, Gu B, Zhu L, Chen C. Mini-midvastus versus mini-medial parapatellar approach in total knee arthroplasty: a prospective, randomized study. Arch Orthop Trauma Surg. 2013 Mar;133(3):389-95. doi: 10.1007/s00402-012-1645-x. Epub 2012 Dec 11. PMID 23229457
- [Background] Nestor BJ, Toulson CE, Backus SI, Lyman SL, Foote KL, Windsor RE. Mini-midvastus vs standard medial parapatellar approach: a prospective, randomized, double-blinded study in patients undergoing bilateral total knee arthroplasty. J Arthroplasty. 2010 Sep;25(6 Suppl):5-11, 11.e1. doi: 10.1016/j.arth.2010.04.003. Epub 2010 Jun 11. PMID 20541889
- [Background] Dalury DF, Dennis DA. Mini-incision total knee arthroplasty can increase risk of component malalignment. Clin Orthop Relat Res. 2005 Nov;440:77-81. doi: 10.1097/01.blo.0000185757.17401.7b. PMID 16239787
- [Background] Berend ME, Ritter MA, Meding JB, Faris PM, Keating EM, Redelman R, Faris GW, Davis KE. Tibial component failure mechanisms in total knee arthroplasty. Clin Orthop Relat Res. 2004 Nov;(428):26-34. doi: 10.1097/01.blo.0000148578.22729.0e. PMID 15534515
- [Background] King J, Stamper DL, Schaad DC, Leopold SS. Minimally invasive total knee arthroplasty compared with traditional total knee arthroplasty. Assessment of the learning curve and the postoperative recuperative period. J Bone Joint Surg Am. 2007 Jul;89(7):1497-503. doi: 10.2106/JBJS.F.00867. PMID 17606788
- [Background] Zhang Z, Gu B, Zhu W, Zhu L, Li Q, Du Y. Minimal invasive and computer-assisted total knee replacement compared with the minimal invasive technique: a prospective, randomized trial with short-term outcomes. Arch Orthop Trauma Surg. 2014 Jan;134(1):65-71. doi: 10.1007/s00402-013-1879-2. Epub 2013 Nov 8. PMID 24202408
- [Background] Seon JK, Song EK, Yoon TR, Park SJ, Bae BH, Cho SG. Comparison of functional results with navigation-assisted minimally invasive and conventional techniques in bilateral total knee arthroplasty. Comput Aided Surg. 2007 May;12(3):189-93. doi: 10.3109/10929080701311861. PMID 17538792
- [Background] Dutton AQ, Yeo SJ, Yang KY, Lo NN, Chia KU, Chong HC. Computer-assisted minimally invasive total knee arthroplasty compared with standard total knee arthroplasty. A prospective, randomized study. J Bone Joint Surg Am. 2008 Jan;90(1):2-9. doi: 10.2106/JBJS.F.01148. PMID 18171951
- [Background] Luring C, Beckmann J, Haibock P, Perlick L, Grifka J, Tingart M. Minimal invasive and computer assisted total knee replacement compared with the conventional technique: a prospective, randomised trial. Knee Surg Sports Traumatol Arthrosc. 2008 Oct;16(10):928-34. doi: 10.1007/s00167-008-0582-2. Epub 2008 Jul 17. PMID 18633597
- [Background] Hasegawa M, Yoshida K, Wakabayashi H, Sudo A. Minimally invasive total knee arthroplasty: comparison of jig-based technique versus computer navigation for clinical and alignment outcome. Knee Surg Sports Traumatol Arthrosc. 2011 Jun;19(6):904-10. doi: 10.1007/s00167-010-1253-7. Epub 2010 Sep 1. PMID 20811732
- [Background] Beldame J, Boisrenoult P, Beaufils P. Pin track induced fractures around computer-assisted TKA. Orthop Traumatol Surg Res. 2010 May;96(3):249-55. doi: 10.1016/j.otsr.2009.12.005. Epub 2010 Apr 8. PMID 20488143
- [Background] Hoke D, Jafari SM, Orozco F, Ong A. Tibial shaft stress fractures resulting from placement of navigation tracker pins. J Arthroplasty. 2011 Apr;26(3):504.e5-8. doi: 10.1016/j.arth.2010.05.009. PMID 20663640
- [Background] Berning ET, Fowler RM. Thermal damage and tracker-pin track infection in computer-navigated total knee arthroplasty. J Arthroplasty. 2011 Sep;26(6):977.e21-4. doi: 10.1016/j.arth.2010.08.012. Epub 2010 Oct 14. PMID 20950996
- [Background] Gulhane S, Holloway I, Bartlett M. A vascular complication in computer navigated total knee arthroplasty. Indian J Orthop. 2013 Jan;47(1):98-100. doi: 10.4103/0019-5413.106927. PMID 23531499
- [Background] Keyes BJ, Markel DC, Meneghini RM. Evaluation of limb alignment, component positioning, and function in primary total knee arthroplasty using a pinless navigation technique compared with conventional methods. J Knee Surg. 2013 Apr;26(2):127-32. doi: 10.1055/s-0032-1319788. Epub 2012 Jul 13. PMID 23288760
- [Background] Chen JY, Chin PL, Tay DK, Chia SL, Lo NN, Yeo SJ. Less outliers in pinless navigation compared with conventional surgery in total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1827-32. doi: 10.1007/s00167-013-2456-5. Epub 2013 Mar 2. PMID 23455388
- [Background] Chen JY, Chin PL, Li Z, Yew AK, Tay DK, Chia SL, Lo NN, Yeo SJ. Radiological outcomes of pinless navigation in total knee arthroplasty: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2015 Dec;23(12):3556-62. doi: 10.1007/s00167-014-3226-8. Epub 2014 Aug 14. PMID 25119055
- [Background] Licini DJ, Meneghini RM. Modern abbreviated computer navigation of the femur reduces blood loss in total knee arthroplasty. J Arthroplasty. 2015 Oct;30(10):1729-32. doi: 10.1016/j.arth.2015.04.020. Epub 2015 Apr 23. PMID 25971778